CLINICAL TRIAL: NCT06534541
Title: Characterizing the Relationships of Genetic Risk and Parental Coercive Feeding Practices With Appetitive Traits and Adiposity Gain Across Early Life.
Brief Title: Genetic Risk, Parental Feeding Practices, and Appetitive Traits in Early Life
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Trustees of Dartmouth College (Other)
Collaborators: Dartmouth-Hitchcock Medical Center (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Dartmouth College (Other)
Responsible Party: Principal Investigator, Jennifer Emond, Associate Professor, Principal Investigator, Trustees of Dartmouth College
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: AWD00012907; 1R01DK136698-01 (NIH)
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Food Cues (Active Comparator): Attentional bias to Food cues experimental measurement
  Interventions: Behavioral: Attentional bias to food cues
- Control Cues (Active Comparator): Attentional bias to food cues control measurement
  Interventions: Behavioral: Attentional bias to food cues

INTERVENTIONS:
Behavioral: Attentional bias to food cues — Measurement of the amount of attention given to food cues

SUMMARY:
The preschool years (2-5 years of age) is a critical timeframe to shape the lifetime risk of obesity. While the causes of obesity are complex, appetitive traits related to overeating, such as high food approach and low food avoidance, are robustly associated with a greater BMI among children. Some children are genetically pre-disposed to expressing obesogenic appetitive traits, and those traits may mediate a genetic risk for obesity. Separately, parental feeding practices are emerging as an important, yet modifiable, influence on children's obesity risk. Coercive control feeding practices, such as strictly limiting a child's intake of highly palatable foods (restriction) and using food to control children's negative emotions (emotional feeding), are believed to be detrimental for young children because they impede self-regulatory skills around eating and may increase the saliency of highly palatable foods. The goal for this project is to disentangle the inter-relationships between coercive control feeding practices, children's obesogenic appetitive traits, and children's dietary intake across the preschool years to understand how coercive control feeding practices ultimately impact children's adiposity gain over time. Importantly, the investigators aim to understand how those effects differ based on children's underlying genetic risk for obesity. The investigators hypothesize that parents will respond to children's obesogenic appetitive traits by exhibiting more coercive control feeding practices (restriction, emotional feeding), which in turn, will promote future increase in obesogenic appetitive traits and overconsumption, leading to excess adiposity gain among children. Importantly, the investigators hypothesize children with a high genetic risk for obesity will be most susceptible to the negative effects of coercive control feeding practices because food is highly salient for them. The investigators will test the hypotheses among a cohort of children aged 2.5 years old using a longitudinal study design with repeated assessments every 6 months until children are 5 years old. If successful, study findings may be leveraged to develop tailored strategies to help parents support healthy eating behaviors among their young children that consider the heterogeneity in obesogenic appetitive traits among young children due to genetic risk factors.

DETAILED DESCRIPTION:
The goal for this project is to disentangle the inter-relationships between coercive control feeding practices, children's obesogenic appetitive traits, and children's dietary intake across the preschool years to understand how coercive control feeding practices ultimately impact children's adiposity gain over time.

The investigators will assess children's genetic risk for obesity via candidate single-nucleotide polymorphisms (SNPs) and a polygenic risk score. Importantly, this novel approach expands upon previous research by including the investigator's lab's proven, objective paradigm to measure children's food approach and overconsumption. Specifically, the investigators will use eye-tracking to measure children's attentional bias to food, an objective metric of food approach. The investigators also include an eating in the absence of hunger paradigm to objectively measure children's overconsumption.

The investigators will test this hypotheses among a cohort of children aged 2.5 years old using a longitudinal study design with repeated assessments every 6 months until children are 5 years old.

ELIGIBILITY:
Inclusion Criteria:

* parent must be ≥18 years old, have primary custody of their child for ≥75% of the month, comprehend verbal and written English and not plan to move out of Vermont or New Hampshire during the study timeframe.
* Children must be ≥2.25 and ≤2.99 years old at first visit and have normal or corrected-to-normal vision to enable eye tracking.

Exclusion Criteria:

* Children with any relevant food allergies or dietary restrictions, taking medication or with a medical condition that affects appetite or attention, or with a relative enrolled in the study will be excluded.

Ages: 27 Months to 72 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 330 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Coercive Parental Food Practices | Measured every 6 months from baseline until 2.5 years after baseline.
  Coercive Parental Food Practices will be assessed using the Child Feeding Questionnaire (CFQ) and Parental Feeding Style Questionnaire (PFSQ). The CFQ restriction subscale, with scores for each of 8 items ranging from 1 to 5 (never to always practice the behavior), will be averaged for a single final Restriction score. The 3 items of the emotional feeding domain from the PFSQ, ranging from 1 to 5 (never to always practice the behavior) will be averaged for a single final Emotional Feeding score.
Appetitive Traits | Measured every 6 months from baseline until 2.5 years after baseline.
  Child appetitive traits will be assessed via parent report using the validated Children's Eating Behavior Questionnaire (CEBQ). The CEBQ includes subscales to measure food approach and food avoidance traits. Final scores for each subscale is computed as the average across subscale items and range from 1 to 5 (never to always express that trait).
Eating in the Absence of Hunger. | Measured every 6 months from baseline until 2.5 years after baseline.
  Eating in the Absence of Hunger. Eating in the absence of hunger will be calculated using established methods (Gilbert-Diamond et al., IJO 2017; Fisher & Birch., AM J of Clin Nutr 2002). The pre- and post-weights of each snack items will be used to calculate the number of kCals a child consumed. Increased kCal consumption is evidence of increased eating in the absence of hunger.
Adiposity | Measured every 6 months from baseline until 2.5 years after baseline.
  Adiposity in children will be operationalized as the age- and sex-adjusted BMI z-score. Child height and weight at each assessment will be measured in-person and be used to calculate age and sex-specific BMI z-scores based on WHO child growth charts. If the child is lost to follow up and we cannot obtain in-person measures, we will abstract height and weight from the child's medical records if they consented to that data collection during the baseline visit.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Emond, PhD, Principal Investigator — Dartmouth College; Diane Gilbert-Diamond, ScD, Principal Investigator — Dartmouth College
Locations (1):
- Dartmotuh College, Hanover, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-06-12): https://cdn.clinicaltrials.gov/large-docs/41/NCT06534541/ICF_000.pdf